CLINICAL TRIAL: NCT01491256
Title: Randomized Comparison Multicenter Trial of High Dose Atorvastatin Pre-treatment on Microcirculatory Dysfunction After Drug-ElutIng Stent Implantation in Patients With Acute Coronary Syndrome
Brief Title: Index of Microcirculatory Resistance After Drug-Eluting Stent Implantation With High Dose Atorvastatin Loading
Acronym: RESIST-ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Korean Society of Circulation (Other)
Responsible Party: Principal Investigator, Bong-Ki Lee, Assistance Professor of Medicine, Kangwon National University School of Medicine, The Korean Society of Circulation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RESIST-ACS
Record Dates: First submitted 2011-12-01; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Index of microcirculatory resistance; atorvastatin; drug-eluting stent; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose Atorvastatin (Active Comparator): Arm of pre-procedural high dose atorvastatin loading
  Interventions: Drug: Pre-procedural High dose atorvastatin loading
- Control (Placebo Comparator): No pre-procedural high dose atorvastatin loading
  Interventions: Drug: No pre-procedural high-dose atorvastatin loading

INTERVENTIONS:
Drug: Pre-procedural High dose atorvastatin loading — Atorvastatin 80 mg loading within 24 hours plus 40mg busting within 2 hours before percutaneous coronary intervention
  Other Names: Lipitor (Pfizer)
  Arms: High dose Atorvastatin
Drug: No pre-procedural high-dose atorvastatin loading — atorvastatin 10mg administration within 24 hours before percutaneous coronary intervention
  Other Names: Lipitor (Pfizer)
  Arms: Control

SUMMARY:
Pre-treatment with statins decreased the incidence of cardiac enzyme increase after percutaneous coronary intervention (PCI) and distal embolization suspected to cause post-PCI myocardial damage. This study evaluates the effect of high dose atorvastatin pre-treatment on post-procedural index of microcirculatory resistance (IMR) values that are introduced for assessing the status of the microcirculation.

DETAILED DESCRIPTION:
One hundred patients with non-ST elevation acute coronary syndrome will be randomly assigned to either high dose atorvastatin pre-treatment group(80 mg loading within 24 hours plus 40mg busting within 2 hours before PCI) or control group(atorvastatin 10mg administration within 24 hours before PCI). An intracoronary pressure/temperature sensor-tipped guidewire is used. Thermodilution curves are obtained during maximal hyperemia. The IMR was calculated from the ratio of the mean distal coronary pressure at maximal hyperemia to the inverse of mean hyperemic transit time. Creatine kinase-myocardial band(CK-MB) and CRP level will be measured at baseline and at 12~24 hours after PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Non-ST elevation acute coronary syndrome planed to elective percutaneous coronary intervention

Exclusion Criteria:

* ST elevation myocardial infarction
* Cardiogenic shock
* Congestive heart failure with pulmonary edema
* Severe left ventricular dysfunction (LVEF < 30%)
* History of previous coronary revascularization therapy
* chronic total coronary occlusion
* 3 vessel disease
* Target lesion at distal segments or branches
* Ostial lesion
* Excessive coronary calcification or thrombi
* Elevated transaminase
* Renal dysfunction (serum creatinine > 2.0mg/dL
* History of myopathy
* Contra-indication to anti-platelet therapy
* Not indicated for percutaneous coronary intervention
* Other co-morbidity with life expectancy less than 1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Index of microcirculatory resistance (IMR) | Immediately after percutaneous coronary intervention
  After stent implantation and adjunctive balloon dilatation, final angiogram will be taken. If the final angiogram shows successful results, IMR will be measured and the procedure will be finished.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events (death, myocardial infarction, target vessel failure | 1 year after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Ki Lee, MD, PhD, Principal Investigator — KangWon National University Hospital
Locations (1):
- Kangwon National University Hospital, Chuncheon, South Korea